CLINICAL TRIAL: NCT05630820
Title: Phase 3 Multicenter, Randomized, Double-Blind, Study to Assess the Efficacy and Safety of Treatment With Bepirovirsen in Nucleos(t)Ide Analogue-treated Participants With Chronic Hepatitis B Virus (B-Well 2)
Brief Title: Study of Bepirovirsen in Nucleos(t)Ide Analogue-treated Participants With Chronic Hepatitis B (B-Well 2)
Acronym: B-Well 2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 219288; 2022-002268-53 (EudraCT Number)
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis B; Hepatitis B, Chronic
Keywords: Hepatitis; Chronic Hepatitis; Chronic Hepatitis B; Hepatitis B Virus; hepatitis B virus e-antigen; Bepirovirsen; Nucleos(t)ide analog; Antisense Oligonucleotide; 202009; 219288; Nucleos(t)ide analogue
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis; Hepatitis, Chronic; Hepatitis B

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double blinded study in which investigators/site staff and the Sponsor will remain blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bepirovirsen (Experimental)
  Interventions: Drug: Bepirovirsen
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bepirovirsen — Bepirovirsen will be administered.
  Arms: Bepirovirsen
Other: Placebo — Matching placebo will be administered.
  Arms: Placebo

SUMMARY:
This study is intended to confirm the efficacy, safety, pharmacokinetic (PK) profile, and the durability of hepatitis B virus surface antigen (HBsAg) suppression observed with bepirovirsen for 24 weeks (with loading doses) as compared to the placebo arm. This study will have 4 stages: a) Double-blind treatment (bepirovirsen or placebo) for 24 weeks. b) Nucleos(t)ide analogue (NA) treatment for 24 weeks. c) NA cessation stage OR Continue NA for 24 weeks. d) Durability of response and follow up for further 24 weeks for participants who stopped NA treatment at Week 48. The arms will be stratified based on HBsAg level (HBsAg greater than or equal to [≥] 100 international unit per milliliter [IU/mL] to less than or equal [≤]1000 IU/mL or greater than [>] 1000 IU/mL to ≤3000 IU/mL) at screening. The total duration of the study, including screening (up to 60 days), the double-blind treatment stage (24 weeks), the On NA only stage (24 weeks), and the NA cessation and durability stages (48 weeks) is up to approximately 104 weeks at maximum for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have documented chronic HBV infection ≥6 months prior to screening and currently receiving stable NA therapy defined as no changes to their NA regimen from at least 6 months prior to Screening and with no planned changes to the stable regimen over the duration of the study.
* Plasma or serum HBsAg concentration >100 IU/mL, but no greater than ≤3000 IU/mL.
* Plasma or serum HBV DNA concentration must be adequately suppressed, defined as plasma or serum HBV DNA <90 IU/mL.
* Alanine aminotransferase (ALT) ≤2 × upper limit of normal (ULN).
* Participants who are willing and able to cease their NA treatment in accordance with the protocol.

Exclusion Criteria:

* Clinically significant abnormalities, aside from chronic HBV infection in medical history (e.g., moderate severe liver disease other than chronic HBV, acute coronary syndrome within 6 months of screening, major surgery within 3 months of screening, significant/unstable cardiac disease, uncontrolled diabetes, bleeding diathesis or coagulopathy) or physical examination.

Co-infection with:

a) Current history of Hepatitis C infection or participants that have been cured for <12 months at the time of screening b) Human immunodeficiency virus (HIV), c) Hepatitis D virus.

* History of or suspected liver cirrhosis and/or evidence of cirrhosis.
* Diagnosed or suspected hepatocellular carcinoma.
* History of malignancy within the past 5 years except for specific cancers that are cured by surgical resection (e.g., skin cancer). Participants under evaluation for possible malignancy are not eligible.
* History of vasculitis or presence of symptoms and signs of potential vasculitis (e.g., vasculitic rash, skin ulceration, repeated blood detected in urine without identified cause) or history/presence of other diseases that may be associated with vasculitis condition (e.g., systemic lupus erythematosus, rheumatoid arthritis, relapsing polychondritis, mononeuritis multiplex).
* History of extrahepatic disorders possibly related to HBV immune conditions (e.g., nephrotic syndrome, any type of glomerulonephritis, polyarteritis nodosa, cryoglobulinemia, uncontrolled hypertension).
* History of alcohol or drug abuse/dependence.
* Currently taking, or took within 3 months of screening, any immunosuppressing drugs (e.g., prednisone), other than a short course of therapy (≤2 weeks) or topical/inhaled steroid use.
* Participants to whom immunosuppressive treatment, including therapeutic doses of steroids is contraindicated, should not be considered for enrolment in the study.
* Currently taking, or has taken within 12 months of Screening, any interferon containing therapy.
* Participants requiring anti coagulation therapies (e.g., warfarin, Factor Xa inhibitors) or anti-platelet agents (like clopidogrel or aspirin) unless treatment can safely be discontinued throughout duration of the study, by the discretion of the investigator. Occasional use is permitted.
* Prior treatment with any oligonucleotide or siRNA within 12 months prior to the first dosing day.
* Prior treatment with bepirovirsen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 857 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants achieving functional cure (FC) with baseline HBsAg ≤3000 IU/mL | Up to 72 weeks
  The number of participants who achieved FC after discontinuation of all chronic HBV treatment (bepirovirsen/placebo and NA) in the absence of rescue medication will be reported. The FC for HBV is defined as Sustained suppression (24 weeks or longer) of HBV DNA <Lower limit of quantification (LLOQ) off all HBV treatment and HBsAg not detected with or without HBsAb after a finite duration of therapy.

SECONDARY OUTCOMES:
Number of participants achieving FC with baseline HBsAg ≤1000 IU/mL | Up to 72 weeks
  The number of participants who achieved FC after discontinuation of all chronic HBV treatment (bepirovirsen/placebo and NA) in the absence of rescue medication will be reported. The FC for HBV is defined as Sustained suppression (24 weeks or longer) of HBV DNA (<LLOQ) off all HBV treatment and HBsAb not detected with or without HBsAb after a finite duration of therapy.
Number of participants achieving sustained suppression of HBV DNA (<LLOQ) with baseline HBsAg ≤3000 IU/mL | Up to 72 weeks
  The number of participants who achieved sustained suppression of HBV DNA after discontinuation of all chronic HBV treatment (bepirovirsen/placebo and NA) in the absence of rescue medication will be reported.
Number of participants achieving sustained suppression of HBV DNA (<LLOQ) with baseline HBsAg ≤1000 IU/mL | Up to 72 weeks
  The number of participants who achieved sustained suppression of HBV DNA after discontinuation of all chronic HBV treatment (bepirovirsen/placebo and NA) in the absence of rescue medication will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (151):
- United States (11):
  - GSK Investigational Site, Centreville, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Glen Burnie, Maryland
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Denison, Texas
  - GSK Investigational Site, Seattle, Washington
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Santa Fe
- Australia (4):
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Fitzroy, Victoria
- Brazil (7):
  - GSK Investigational Site, Botucatu
  - GSK Investigational Site, Fortaleza
  - GSK Investigational Site, Nova Iguaçu
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, Vitória
- Bulgaria (4):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sliven
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (6):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
- China (20):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Hefei
  - GSK Investigational Site, Kunming
  - GSK Investigational Site, Liuchow
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shenzhen
  - GSK Investigational Site, Taiyuan
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Ürümqi
  - GSK Investigational Site, Wuhan
  - GSK Investigational Site, Xi'an
  - GSK Investigational Site, Xiamen
  - GSK Investigational Site, Zhengzhou
  - GSK Investigational Site, Zunyi
- France (7):
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Toulouse
- Germany (3):
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion Crete
  - GSK Investigational Site, Thessaloniki
- Hungary (3):
  - GSK Investigational Site, Szeged
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Zalaegerszeg
- India (11):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Kanpur
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Raipur
  - GSK Investigational Site, Secunderabad
- Italy (8):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Sassari
  - GSK Investigational Site, Torino
- Japan (13):
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamaguchi
  - GSK Investigational Site, Yamanashi
- Malaysia (6):
  - GSK Investigational Site, Johor Bahru
  - GSK Investigational Site, Kota Bharu Kelantan
  - GSK Investigational Site, Kota Kinabalu
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kuala Terengganu
  - GSK Investigational Site, Kuantan
- GSK Investigational Site, Aguascalientes, Mexico
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Papatoetoe Auckland
- GSK Investigational Site, Panama City, Panama
- Philippines (4):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Makati City
  - GSK Investigational Site, Pasig
  - GSK Investigational Site, Silang
- Poland (3):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Mysłowice
  - GSK Investigational Site, Żychlin
- Romania (5):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Galati
  - GSK Investigational Site, Oradea
- South Korea (5):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Ulsan
- Spain (9):
  - GSK Investigational Site, Alcorcon Madrid
  - GSK Investigational Site, Badajoz
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Sabadell Barcelona
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Zaragoza
- Taiwan (4):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- GSK Investigational Site, Chiang Mai, Thailand
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Izmir
- United Kingdom (4):
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Middlesbrough
  - GSK Investigational Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/